CLINICAL TRIAL: NCT07274462
Title: A Randomized Controlled Study of Daratumumab for Microvascular Inflammation (MVI) in Kidney Transplant Recipients With or Without Donor-Specific Antibodies
Brief Title: DARA-MVI Study (Daratumumab for Microvascular Inflammation in Kidney Transplantation)
Acronym: DARA-MVI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Martin (Other)
Responsible Party: Principal Investigator, Matej Vnucak, associate professor, University Hospital, Martin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TNO DARA MVI
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Microvascular Inflammation - MVI in Kindey Transplant Recipients
Keywords: Kidney transplantation; Microvascular inflammation; acute rejection
MeSH Terms: interventions — daratumumab; Observation; Standard of Care

STUDY DESIGN:
Masking Description: Open-label (pathology and laboratory assessments blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Daratumumab (Darzalex®) (Experimental): Participants with biopsy-proven microvascular inflammation (MVI) (Banff g ≥1 and/or ptc ≥1), C4d-negative, randomized to receive daratumumab 1800 mg SC once monthly for 3 months, in addition to standard post-transplant care and monitoring (DSA, dd-cfDNA, eGFR).
  Interventions: Drug: DARATUMUMAB (DARZALEX®)
- Active Comparator: Observation (Standard Care) (Active Comparator): Participants with biopsy-proven MVI, C4d-negative, randomized to observation under standard post-transplant care and monitoring (DSA, dd-cfDNA, eGFR) without daratumumab treatment.
  Interventions: Other: Observation (Standard Care)

INTERVENTIONS:
Drug: DARATUMUMAB (DARZALEX®) — Daratumumab 1800 mg subcutaneously once monthly × 3 doses plus standard monitoring of DSA and dd-cfDNA every 3 months.
  Other Names: Experimental: Daratumumab (Darzalex®)
  Arms: Experimental: Daratumumab (Darzalex®)
Other: Observation (Standard Care) — Standard post-transplant management and monitoring per institutional protocol. Includes serial measurement of DSA and donor-derived cell-free DNA every 3 months, eGFR monitoring, and repeat biopsy at 12 months.
  Other Names: Active Comparator: Observation (Standard Care)
  Arms: Active Comparator: Observation (Standard Care)

SUMMARY:
The DARA-MVI Study is a prospective, randomized, controlled, open-label trial designed to evaluate the effect of daratumumab on microvascular inflammation (MVI) in kidney transplant recipients with C4d-negative biopsies. Participants with biopsy-proven MVI will be randomized to receive either daratumumab or observation with standard monitoring. The study will assess changes in histologic MVI score, donor-derived cell-free DNA (dd-cfDNA), donor-specific antibodies (DSA), and graft function over 12 months.

DETAILED DESCRIPTION:
Microvascular inflammation (MVI) is a histologic feature associated with antibody-mediated injury and poor long-term graft outcomes in kidney transplantation. However, the optimal management of MVI-particularly in C4d-negative, donor-specific antibody (DSA)-negative cases-remains undefined. Recent data suggest that activation of plasma cells and long-lived memory B cells may contribute to persistent endothelial injury even in the absence of circulating DSA.

Daratumumab, a human monoclonal antibody targeting CD38, has demonstrated potent depletion of plasma cells and immunomodulatory effects in autoimmune diseases and in early reports of antibody-mediated rejection (ABMR) resistant to standard therapy. Building on this evidence, the DARA-MVI study aims to evaluate whether daratumumab can attenuate microvascular inflammation and stabilize graft function in kidney transplant recipients with biopsy-proven MVI but negative C4d staining.

This is a prospective, randomized, open-label, controlled trial enrolling adult kidney transplant recipients who undergo indication or surveillance biopsy revealing MVI (glomerulitis [g] and/or peritubular capillaritis [ptc] ≥ 1). Participants will be randomized in a 1:1 ratio to receive either (1) daratumumab subcutaneous therapy (1800 mg monthly for 3 months) or (2) observation under standard clinical monitoring. A non-randomized reference group of biopsy-negative, DSA-negative, and dd-cfDNA-negative transplant recipients will serve as a comparative baseline for biomarker trajectories.

All participants will undergo structured follow-up for 12 months, including serial assessment of graft function, dd-cfDNA (fraction and copy number), and DSA at baseline and every 3 months. Repeat biopsy at 12 months will evaluate histologic response (change in Banff MVI score: g + ptc).

The primary objective is to determine whether daratumumab reduces microvascular inflammation compared to observation. Secondary objectives include evaluation of changes in donor-derived cell-free DNA, emergence or resolution of DSA, estimated glomerular filtration rate (eGFR), and safety outcomes (adverse events, infection, and cytopenia).

The study also aims to explore correlations between histologic, molecular (dd-cfDNA), and serologic (DSA) indicators of alloimmune activity. This will help determine whether daratumumab can interrupt subclinical alloimmune injury and delay chronic graft deterioration.

If successful, this study could define a novel therapeutic approach for antibody-independent microvascular inflammation and clarify the role of plasma-cell-directed therapies in complex post-transplant immune responses.

ELIGIBILITY:
Inclusion:

Age ≥ 18, kidney transplant recipients (first or higher, living or deceased donor), biopsy-proven MVI (g ≥ 1 and/or ptc ≥ 1), C4d-negative, DSA-negative (Cohort 1) or DSA-positive (Cohort 2), informed consent.

Exclusion:

C4d-positive biopsy, active TCMR ≥ IA, infection or malignancy, multi-organ transplant, prior anti-CD38 therapy, pregnancy, breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Change in microvascular inflammation score (Banff g + ptc) between baseline and 12 months. | Baseline (study entry) and 12 months after randomization
  The composite microvascular inflammation (MVI) score, defined as the sum of glomerulitis (g) and peritubular capillaritis (ptc) scores according to the Banff classification (range 0-6), will be assessed on kidney-allograft biopsy specimens obtained at baseline and at 12 months. The change in total MVI score (ΔMVI = [g + ptc]₁₂ₘ - [g + ptc]₀) will be compared between treatment arms to evaluate the effect of daratumumab on microvascular inflammation.

CONTACTS AND LOCATIONS:
Locations (1):
- Transplant-nephrology department, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the published results will be made available upon reasonable request from qualified researchers after publication, following institutional and ethical approval. Supporting documents (protocol, statistical analysis plan) may also be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 01/MAR/2025 for 20 years

DOCUMENTS (1):
  • Study Protocol (2025-11-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT07274462/Prot_000.pdf